CLINICAL TRIAL: NCT05967507
Title: Laryngoscopy for Neonatal and Infant Airway Management with Supplemental Oxygen At Different Flow Rates (OPTIMISE-2): a Multi-center, Non-inferiority, Prospective Randomized Controlled Trial
Brief Title: Laryngoscopy for Neonatal and Infant Airway Management with Supplemental Oxygen At Different Flow Rates (OPTIMISE-2)
Acronym: OPTIMISE-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thomas Riva (Other)
Collaborators: University Hospital, Geneva (Other); Kantonsspital Aarau (Other); Centre Hospitalier Universitaire Vaudois (Other); Charite University, Berlin, Germany (Other); Royal Perth Hospital (Other); The Hospital for Sick Children (Other); Istituto Giannina Gaslini (Other)
Responsible Party: Sponsor-Investigator, Thomas Riva, Prof. Dr. med., Insel Gruppe AG, University Hospital Bern
Organization: Insel Gruppe AG, University Hospital Bern (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OPTIMISE-2-trial
Record Dates: First submitted 2023-07-19; First posted 2023-08-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-01

CONDITIONS: Airway Management

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): 0.2 L/kg/min FiO2 1.0 low-flow nasal supplemental oxygen with conventional nasal cannula during tracheal intubation performed with the C-MAC videolaryngoscope (Karl Storz, Tuttlingen, Germany) with Miller-blade or Macintosh-blade size No. 0 or No. 1.
  Interventions: Device: Low-flow nasal supplemental oxygen with a conventional nasal cannula during tracheal intubation with the C-MAC video laryngoscope
- Control group (Active Comparator): 2 L/kg/min FiO2 1.0 high-flow nasal supplemental oxygen with the Optiflow (Fisher & Paykel Healthcare, Auckland, New Zealand) during tracheal intubation performed with the C-MAC videolaryngoscope (Karl Storz, Tuttlingen, Germany) with Miller-blade or Macintosh-blade size No. 0 or No. 1.
  Interventions: Device: High-flow nasal supplemental oxygen (Fisher & Paykel, Auckland, New Zealand) during tracheal intubation with the C-MAC video laryngoscope

INTERVENTIONS:
Device: Low-flow nasal supplemental oxygen with a conventional nasal cannula during tracheal intubation with the C-MAC video laryngoscope — 0.2 L/kg/min FiO2 1.0 low-flow nasal supplemental oxygen with a conventional nasal cannula during tracheal intubation with the C-MAC video laryngoscope (Karl Storz, Tuttlingen, Germany) with Miller-blade or Macintosh-blade size No. 0 or No. 1.
  Arms: Intervention group
Device: High-flow nasal supplemental oxygen (Fisher & Paykel, Auckland, New Zealand) during tracheal intubation with the C-MAC video laryngoscope — 2 L/kg/min FiO2 1.0 high-flow nasal supplemental oxygen (Fisher & Paykel, Auckland, New Zealand) during tracheal intubation with the C-MAC video laryngoscope (Karl Storz, Tuttlingen, Germany) with Miller-blade or Macintosh-blade size No. 0 or No. 1.
  Arms: Control group

SUMMARY:
This study aims to investigate the optimal oxygen flow rate needed during tracheal intubation with the C-MAC video laryngoscope (Karl Storz, Tuttlingen, Germany) using Miller-blade or Macintosh-blade size No. 0 or No. 1 in the operating room or intensive care unit. The investigators hypothesize that the difference between low-flow and high-flow supplemental oxygen is negligible.

DETAILED DESCRIPTION:
Eligible children will be prepared for intubation according to the local SOPs of the pediatric anesthesia departments. Mandatory monitoring will consist of: SpO2, HR, NIBP.

Induction of anesthesia: If feasible, all children included in this protocol will be pre-oxygenated before induction of anesthesia for one minute through face-mask with FiO2 1.0 and flow rates of 6-10L/min. The induction of anesthesia for tracheal intubation will be performed using a combination of sedative/hypnotic drugs, opioids and non-depolarizing muscle relaxant.

The following medications will be mandatory as per protocol:

* A neuromuscular blocking agent (NMBA): Rocuronium 0.5-1 mg/kg, Cis-Atracurium 0.2-0.5 mg/kg, Atracurium 0,5 mg/kg, Vecuronium 0.1 mg/kg, Mivacurium 0.2 - 0.3 mg/kg or Succinylcholine 2 mg/kg.
* One or more of the following hypnotic agents (Thiopentone 4-7 mg/kg, Ketamine 0.5-2 mg/kg, Propofol 1-4 mg/kg, Midazolam 0.5-1 mg/kg, Sevoflurane up to 8%).
* An opioid drug and anticholinergic can be chosen and administered at the discretion of the anesthetist in charge.

Before intubation: After induction of anesthesia and the administration of a NMBA, bag-mask ventilation with FiO2 1.0 (flow rates of 6-10 L/min) will be performed for 60 seconds until apnea sets in. After induction all patients will be paralyzed to facilitate airway management. Full neuromuscular blockade will be assessed by train-of-four (TOF) monitoring. Thereafter oxygen administration, laryngoscopy and tracheal intubation are performed.

During intubation: The administration of oxygen during intubation is mandatory for every study participant and is randomized as follows:

Low-flow Oxygen Group: For orally intubated children, the administration of low-flow oxygen (0.2 L/kg/min FiO2 1.0) takes place via conventional nasal cannula (Intersurgical, Wokingham, UK). For nasally intubated children, the administration of low-flow oxygen (0.2 L/kg/min FiO2 1.0) takes place via a nasal oxygen sponge cannula (Vygon, Ecouen, France) adapted to the dimension of nare. After administration of low-flow oxygen laryngoscopy and tracheal intubation are performed.

High-Flow Oxygen Group (control-group): For all orally intubated children, the administration of high-flow oxygen (2 L/kg/min FiO2 1.0) takes place via nasal cannula with the Optiflow (Fisher & Paykel Healthcare, Auckland, New Zealand). For nasally intubated children, the administration of low-flow oxygen (2 L/kg/min FiO2 1.0) takes place via the anaesthesia circuit through the tracheal tube placed in the nose. After administration of high-flow oxygen laryngoscopy and tracheal intubation are performed.

For a premature neonate < 1kg an uncuffed tube ID 2.5 will be used. For premature babies and newborn between 1kg and 3.0 kg an uncuffed tube ID 3.0 will be used. For babies > 3.0 kg - 8 months a cuffed tube ID 3.0 or an uncuffed tube 3.5 will be used. For infants 8 months - 12 months a cuffed tube ID 3.5 or an uncuffed tube 4.0 will be used. Based on the group of randomization, the child will receive supplemental oxygen low-flow via a conventional nasal cannula vs high-flow with the Optiflow (Fisher & Paykel Healthcare, Auckland, New Zealand).

Miller-blade or Macintosh-blade size No. 0 will be used for children < 1 kg. In cases of unexpected difficult intubation, the difficult airway algorithm (18) will be followed. After the first unsuccessful intubation attempt with the randomized flowrate, the investigators encourage to perform a second attempt with the same rate but based on the clinical judgment the intubating physician can proceed to an attempt with the same technique, or change the flow rate, blade size or the type of laryngoscope. A maximum of 4 intubation attempts in total will be performed. The last intubation attempt must be performed by the most experienced physician in the room. Additional devices like stylet, bougie, etc., can be used at any stage of the intubation process. If the intubation remains unsuccessful the difficult airway algorithm will be followed (Appendix) and a supraglottic airway - SGA will be inserted.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients requiring oral or nasal tracheal intubation for elective, semi-elective, or urgent surgical and non-surgical indications.
* Neonates and infants up to 52 weeks postconceptual age, with legal guardians providing written informed consent before the intervention

Exclusion Criteria:

* Prediction of difficult intubation upon physical examination or previous history of difficult intubation, mandating a technique different than direct laryngoscopy to secure the airway;
* Congenital heart disease demanding FiO2 < 1.0
* Cardiopulmonary collapse requiring advanced life support
* Intubation for emergency surgical and non-surgical indications.

Max Age: 52 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1192 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
First attempt success rate | 15 minutes
  The primary study outcome is to evaluate the first attempt success rate of oral and nasal tracheal intubation with the C-MAC video laryngoscope (Karl Storz, Tuttlingen, Germany) with supplemental oxygen with low-flow vs high flow among neonates and infants up to 52 weeks postconceptual age. A successful tracheal intubation (ETI) attempt is defined as successful placement of a tracheal tube in the trachea, confirmed by visualization of the tube passing the vocal cords, a waveform capnography suggesting correct ETT placement and auscultation of breath sounds in the lungs.

SECONDARY OUTCOMES:
Occurrence of severe desaturation | 15 minutes
  Occurrence and duration of moderate and severe desaturation (SpO2 < 10% and SpO2 < 20% from baseline), with or without bradycardia, during intubation.
Overall number of intubation attempts | 15 minutes
  Overall number of intubation attempts
First attempt success rate of tracheal intubation | 15 Minutes
  First attempt success rate of tracheal intubation
Time required for intubation | 5 minutes
  Time required for intubation (in seconds, defined from the first introduction of laryngoscope between the lips till successful lung ventilation defined as positive capnography)
First EtCO2 after successful intubation | 10 minutes
  Value in mmHg or kPa of the first reliable etCO2 reading after successful intubation
Cormack-Lehane score | 5 minutes
  Cormack-Lehane score at any attempt of laryngoscopy
The need for additional devices | 5 minutes
  The need for additional devices used at any step of intubation
Respiratory complications | 24 hours
  Respiratory complications or complications of airway management within the first 24 hours, such as airway injury, cardiopulmonary resuscitation, bleeding, aspiration of gastric contents, post-extubation stridor, laryngospasm, bronchospasm, need for High Flow Nasal Oxygen (if not preoperatively on oxygen), need for low flow nasal oxygen (if not preoperatively on oxygen) or need for re-intubation will be recorded. Respiratory complications are defined as the need for re-intubation after being extubated, persistent stridor (even if oxygen is not required), respiratory failure, the occurrence of pneumothorax or the need for any additional diagnostic examination following respiratory problems (i.e., bronchoscopy, radiology).
Duration of severe desaturation | 15 minutes
  Duration of moderate and severe desaturation (SpO2 < 80%), with or without bradycardia, during intubation.
Percentage of Glottic Opening (POGO) score | 5 minutes
  Percentage of Glottic Opening (POGO) score at any attempt of laryngoscopy, (0-100%). 100% best glottic opening

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Riva, MD, Study Chair — University of Bern
Locations (6):
- Canada (2):
  - Dept. Anesthesia, The Hospital for Sick Children, Toronto, Ontario
  - Dept. Anesthesia, Montreal Children's Hospital, McGill University Health Centre, Montreal
- Germany (2):
  - Deutsches Herzzentrum der Charité and Charité, Berlin
  - Department of Cardiac Anesthesiology and Intensive Care Medicine, Charité Universitätsmedizin, Berlin
- Switzerland (2):
  - Inselspital, Bern, Canton of Bern
  - CHUV Centre Hospitalier Universitaire Vaudois, Lausanne

IPD SHARING:
Plan to Share IPD: No